CLINICAL TRIAL: NCT05113758
Title: "SARCOPENIA MEASURED BY ULTRASOUND IN HOSPITALIZED OLDER ADULTS" (ECOSARC Study).
Brief Title: Sarcopenia Measured by Ultrasound in Hospitalized Older Adults
Acronym: ECOSARC
Status: Completed | Type: Observational
Sponsor: Pedro Abizanda (Other)
Collaborators: Hospital Universitario Getafe (Other); Hospital Infanta Sofia (Other); Hospital Universitario Infanta Leonor (Other); Hospital Universitario La Paz (Other); Puerta de Hierro University Hospital (Other); Hospital Virgen del Valle de Toledo (Unknown)
Responsible Party: Sponsor-Investigator, Pedro Abizanda, Principal Investigator, Complejo Hospitalario Universitario de Albacete
Organization: Complejo Hospitalario Universitario de Albacete (Other)
Other Study IDs: ABZ-ECO-2018-01
Record Dates: First submitted 2021-10-29; First posted 2021-11-09 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Sarcopenia
Keywords: sarcopenia; ultrasound; aged; hospitalized
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: muscle ultrasound — All participants will undergo a muscle ultrasound on admission and at discharge

SUMMARY:
Observational prospective study in older adults admitted to an Acute Geriatric Unit, in which sarcopenia will be evaluated by ultrasound in the anterior rectus femoris muscle.

DETAILED DESCRIPTION:
The main objective of the study is to estimate, by means of portable ultrasound, parameters of muscle quantity and quality (anterior rectus femoris muscle area, width and echostructure ) in older adults hospitalized in Acute Geriatric Units for medical reasons.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 69 years of age.
* Hospitalization for a medical cause in Acute Geriatric Units.
* Holden's Functional Ambulation Classification Scale at level 1 or higher.
* Informed consent signed by the patient or legal representative.

Exclusion Criteria:

* Terminal condition or life expectancy of less than 6 months.
* Impossibility or refusal to undergo muscle ultrasound.
* Refusal for follow-up
* Severe dementia stage Global Deteriorating Scale: 7
* Impossibility in the opinion of the investigators to complete the necessary data for the study.

Min Age: 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients over 69 years of age admitted to Acute Geriatric Units.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of sarcopenia on admission | 72 hours
  Prevalence of sarcopenia on admission. A prevalent case of sarcopenia will be considered if a patient fulfills the EWGSOP2 at admission
Incidence of sarcopenia between admission and discharge | 15 days
  An incident case of sarcopenia will be considered if a patient not fulfilling EWGSOP2 diagnostic criteria on admission, will meet diagnostic criteria at discharge of sarcopenia at discharge (diagnosis will be considered as a dichotomous variable -yes/no-).
Muscle mass (the anterior rectus femoris muscle) | 15 days
  The evolution of muscle mass between admission and discharge will be assessed by ultrasound

SECONDARY OUTCOMES:
Minimal nutritional assessment (MNA-SF) score | 72 hours
  The mini-nutritional assessment - short form is a simple, non - invasive and validated scale for the detection of malnutrition in older adults. It takes into account the patient's loss of appetite, weight loss, motor skills, recent health status, neuropsychological disorders. The maximum score of the MNA-SF is 14:
  Greater than or equal to 11: normal nutritional status. Between 8 and 11: risk of malnutrition. Less than 8: malnutrition.
Hand grip strength | 15 days
  Using a hand-held dynamometer
4-meter walking speed test | 15 days
  The evolution of the value of the 4-meter walking speed test between admission and discharge will be assessed.
ADL (Activities of Daily Living) questionnaire | 3 months
  the ADL questionnaire will also be performed on admission, at discharge, and at 3 months.
SPPB score (SHORT PHYSICAL PERFORMANCE BATTERY score) | 15 days
  Short Physical Performance Battery (SPPB): score range 0-12, higher score means a better outcome
Mortality | 3 months
  Mortality will be measured with vital status at 3 months.
Length of stay, days | 15 days
  Day of admission to day of discharge
Readmission(s) after index hospitalization | 3 months
  Readmission(s) after index hospitalization, Dichotomous outcome (yes/no)
Emergency department (ED) visit(s) | 3 months
  ED visit(s) after index hospitalization, Dichotomous outcome (yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Abizanda, MD, PhD, Principal Investigator — Complejo Hospitalario Universitario de Albacete (SESCAM)
Locations (1):
- Complejo Hospitalario Universitario de Albacete, Albacete, Spain

REFERENCES:
- [Derived] Lopez Jimenez E, Neira Alvarez M, Menendez Colino R, Checa Lopez M, Grau Jimenez C, Perez Rodriguez P, Vasquez Brolen B, Arias Munana E, Ramirez Martin R, Alonso Bouzon C, Amor Andres MS, Bermejo Boixareu C, Branas F, Alcantud Ibanez M, Alcantud Corcoles R, Cortes Zamora EB, Gomez Jimenez E, Romero Rizos L, Avendano Cespedes A, Hernandez Socorro CR, Abizanda P. Muscle mass loss measured with portable ultrasound in hospitalized older adults: The ECOSARC study. J Nutr Health Aging. 2024 Jan;28(1):100010. doi: 10.1016/j.jnha.2023.100010. Epub 2023 Dec 14. PMID 38267149
- [Derived] Lopez Jimenez E, Neira Alvarez M, Ramirez Martin R, Alonso Bouzon C, Amor Andres MS, Bermejo Boixareu C, Branas F, Menendez Colino R, Arias Munana E, Checa Lopez M, Grau Jimenez C, Perez Rodriguez P, Alcantud Ibanez M, Vasquez Brolen B, Oliva J, Pena Longobardo LM, Alcantud Corcoles R, Cortes Zamora EB, Gomez Jimenez E, Romero Rizos L, Avendano Cespedes A, Hernandez Socorro CR, Abizanda P. "SARCOPENIA MEASURED BY ULTRASOUND IN HOSPITALIZED OLDER ADULTS" (ECOSARC): multi-centre, prospective observational study protocol. BMC Geriatr. 2023 Mar 22;23(1):163. doi: 10.1186/s12877-023-03891-5. PMID 36949412